CLINICAL TRIAL: NCT02055638
Title: An Exploratory Phase II Study to Determine the Safety, Tolerability and Activity of a Novel Vasopressin 1a Receptor Antagonist (SRX246) in Adults With Diagnostic and Statistical Manual Version 5 (DSM-5) Intermittent Explosive Disorder (IED)
Brief Title: Safety, Tolerability and Activity of SRX246 in Adults With Intermittent Explosive Disorder
Acronym: AVN009
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Azevan Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AVN009
Record Dates: First submitted 2014-02-03; First posted 2014-02-05 (Estimated); Results first posted 2019-10-29 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Intermittent Explosive Disorder
Keywords: Intermittent Explosive Disorder; IED; Aggression; SRX246; Vasopressin 1a Receptor Antagonist; V1a
MeSH Terms: conditions — Disruptive, Impulse Control, and Conduct Disorders; Aggression | interventions — SRX246

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SRX246 (Experimental): SRX246 capsules, 120mg bid for 4 weeks followed by 160mg bid for 4 weeks
  Interventions: Drug: SRX246
- Placebo (Placebo Comparator): Placebo capsules to match the amount of SRX246 capsules for 8 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SRX246 — capsules
  Arms: SRX246
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study is designed to explore the safety and tolerability, and to compare the activity of SRX246 against placebo, in adults with Intermittent Explosive Disorder (IED).

Adult Male and Female subjects with a current diagnosis of IED will be enrolled. After a two-week baseline lead-in phase, study subjects who continue to meet enrollment criteria will be randomized to either SRX246 or Placebo treatment groups.

Study subjects will be examined and asked to answer questionnaires at weekly scheduled visits throughout the trial. The study results will be determined based on any changes observed over the study period.

DETAILED DESCRIPTION:
This exploratory Phase II study has been designed to examine the safety and tolerability profile, and to compare the activity of the novel V1a vasopressin antagonist (SRX246) against placebo, in adults with DSM-5 Intermittent Explosive Disorder (IED).

Adult Male and Female subjects with a current DSM-5 diagnosis of IED will be enrolled. All subjects will undergo systematic diagnostic assessment for DSM-5 Axis I and II disorders. Subjects with DSM-5 IED (without current, co-morbid, DSM-5 Major Depression) whose: (a) Life History of Aggression (LHA) score is > 12, (b) Overt Aggression Scale Modified (OAS-M) "Irritability" score is > 6 and, (c) screening OAS-M "Aggression" score is > 15, will be entered into a two-week baseline lead-in phase.

After the lead-in phase, study subjects who continue to meet OAS-M criteria will be randomized to one of the two (2) treatment conditions and stratified by gender so that equal numbers of males and females are assigned to SRX246 and Placebo Groups. Those who do not meet the criteria will exit the protocol at that time. Treatment Conditions: (a) 8-week course of SRX246 (4 weeks at 120 mg bid, and 4 weeks at 160 mg bid) or (b) 8-week course of Placebo, followed by a one-week "taper" to withdraw subjects from study medication.

IED subjects in all conditions will have structured diagnostic interview sessions and questionnaires administered throughout the trial. Blinding to treatment condition will be maintained by using different personnel for these activities. Analysis of a change from baseline in the diagnostic measures will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female (Women of child bearing potential must be non-pregnant, non-lactating and agree to be on an acceptable method of contraception.)
* Age 21 to 55 years, inclusive.
* In good general physical health as determined by medical history, a baseline physical examination, vital signs, clinical laboratory tests and electrocardiogram (EKG) measurement.
* Current IED by DSM-5
* LHA-Aggression ≥ 12.
* OAS-M Irritability score ≥ 6, and OAS-M Total Aggression score ≥ 15, respectively at Visit 1
* Mean Irritability and Total Aggression scores for Visit 2 and Visit 3, ≥ 6 and ≥ 15, respectively.
* Subject is willing and able to sign written informed consent prior to receipt of any study medication or beginning study procedures.
* Subject is willing and able to follow instructions, comply with the protocol requirements and make all required study visits.

Exclusion Criteria:

* Subject with a positive test for alcohol and/or drugs of abuse at screening or at any time during the study.
* Presence of any of the following serious and active medical conditions: Seizure Disorder (n.b.: history of < 2 febrile seizures prior to one year of age is acceptable); Demyelinating or Progressive Degenerative Disorders; central nervous system (CNS) Infection; Progressive Degenerative Neurological Disorder; Ischemic Heart Disease, Respiratory Disease, Renal Disease; Liver Disease; Type I Diabetes; Malignant Neoplasm; Hyper- or Hypo-Coagulopathy; Acquired Immuno-Deficiency Syndrome (AIDS).
* Routine or as needed consumption of medications or herbal supplements that the subject is unable or unwilling to discontinue during the study.
* Other ongoing psychotherapeutic treatment for the treatment of IED or anger begun less than three months before entry into this study.
* Not Current DSM-5 IED.
* LHA score < 12 at Visit 1 (screen).
* OAS-M Irritability score < 6 or OAS-M Total Aggression score < 15 at Visit 1 (screen).
* Current major depressive episode or life history of bipolar disorder, schizophrenia, organic mental syndrome, or mental retardation.
* Current DSM-5 Substance Use Disorder of moderate or greater severity (i.e., ≥ 4 Substance Use Disorder (SUD) symptoms).
* Active suicidal ideation as determined by clinical assessment and Columbia-Suicide Severity Rating Scale (C-SSRS).
* Evidence of any out-of range laboratory value at screening that has not been reviewed, approved and documented as not clinically significant by the Study Investigator.
* A history of significant drug allergy or systemic allergic disease (e.g., urticaria, atopic dermatitis), or any known/suspected hypersensitivity to SRX246.
* A general medical or psychological condition or behavior, including current substance dependence or abuse that, in the opinion of the investigator, might not permit the subject to complete the study or sign the informed consent.
* Unwilling/unable to sign informed consent document.
* Any clinically significant abnormality on screening resting 12-lead EKG (e.g., heart block, conduction disorders, ventricular and/or atrial arrhythmias).
* Any other condition or clinically significant abnormal findings on the physical examination, medical history, or clinical laboratory results during screening that, in the opinion of the Study Investigator, would make the subject unsuitable for the study or put them at additional risk.
* Inability to understand or follow study instructions.
* Treatment with an investigational drug within 30 days preceding the first dose of study medication.
* Women who are currently breastfeeding and/or lactating.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 97 (Actual)
Dates: Start 2014-05; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - University of Chicago, Department of Psychiatry, Chicago, Illinois
  - Psychiatric Care and Research Center, O'Fallon, Missouri
  - SPRI Clinical Trials, LLC, Brooklyn, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Lindner Center of HOPE, Mason, Ohio
  - Rhode Island Hospital, Department of Psychiatry, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One additional subject was enrolled than planned, due to timing of screening and notification to sites of ceasing planned enrollment.
Groups:
- Placebo: Placebo capsules to match the amount of SRX246 capsules for 8 weeks
  Placebo
Period: Overall Study
Arm/Group | SRX246 | Placebo
Started | 49 | 48
Completed | 39 | 40
Not Completed | 10 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SRX246 | Placebo | Total
Number analyzed (Participants) | 49 | 48 | 97
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 49 | 48 | 97
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 29 | 28 | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 7
  Not Hispanic or Latino | 45 | 43 | 88
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 29 | 31 | 60
  White | 16 | 12 | 28
  More than one race | 3 | 4 | 7
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 49 | 48 | 97

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability
Description: measured as the number of participants with adverse events
Time Frame: from initial dose of intervention until completion of the study up to 8 weeks
Population: Intent to treat
Measure: Number; unit: participants
Arm/Group | SRX246 | Placebo
Number analyzed (Participants) | 49 | 48
participants
  adverse events (AE) | 28 | 21
  serious adverse events (SAE) | 0 | 0

2. Other Pre Specified Outcome: Overt Aggression Scale Modified (OAS-M) Total Aggression Score
Description: Change from Baseline OAS-M Score. Higher values represent a worse outcome. The OAS-M contains 3 scales: Aggression (Questions [Q]1 to 4), Irritability (Q5 to 6), and Suicidality (Q7 to 7b). Aggression total score was calculated by summing the weighted scores in Q1 to 4. Scores for each question ranged from 0 (no events) to 5 (very severe events). Total scores ranged from 0 (no aggression) to any number with no upper limit depending on the frequency of aggressive behavior in a week.
Time Frame: Comparison of baseline score to score at end of treatment period of 8 weeks
Population: those that took study drug and had sufficient data for analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SRX246 | Placebo
Number analyzed (Participants) | 39 | 41
score on a scale | -29.55 (37.343) | -30.43 (34.082)

ADVERSE EVENTS:
Time Frame: from first dose of study drug to last follow-up visit, up to 8 weeks
Arm/Group | SRX246 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/48
Other Adverse Events (participants affected / at risk) | 9/49 | 7/48
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SRX246 (N=49) | Placebo (N=48)
Headache (Nervous system disorders) | 3 (3) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 2 (2)
Dry Mouth (Gastrointestinal disorders) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No